CLINICAL TRIAL: NCT03961126
Title: Pilot Study of Vulvar Lichen Sclerosus (VLS) Treatment Using Adipose Tissue Associated With Autologous Platelet-rich Plasma (PRP).
Brief Title: Evaluation of Vulvar Lichen Sclerosus Treatment Using Adipose Tissue Associated With Autologous Platelet-rich Plasma.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Instituto de Investigacion Sanitaria La Fe (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LIQUENIA
Record Dates: First submitted 2019-05-17; First posted 2019-05-23 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Vulvar Lichen Sclerosus
Keywords: Vulvar Lichen Sclerosus; Autologous Platelet-rich Plasma (PRP)
MeSH Terms: conditions — Vulvar Lichen Sclerosus | interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group autologous platelet-rich plasma injection (Experimental): Patients will receive 2 separate infiltrations for three months by intra and subdermal injection of autologous fatty tissue (20cc) associated with autologous platelet-rich plasma (4cc) in each half vulvar.
  Interventions: Drug: Injection of autologous fatty tissue associated with autologous platelet-rich plasma.
- Group Control (Active Comparator): Patients will receive a maintenance treatment of topical therapy with corticosteroids (clobetasol 0.05%) that will be administered by usual clinical practice.
  Interventions: Drug: Corticosteroids (clobetasol 0.05%)

INTERVENTIONS:
Drug: Injection of autologous fatty tissue associated with autologous platelet-rich plasma. — Patients will receive 2 separate infiltrations for three months by intra and subdermal injection of autologous fatty tissue (20cc) associated with autologous platelet-rich plasma (4cc) in each half vulvar.
  Other Names: Experimental
  Arms: Group autologous platelet-rich plasma injection
Drug: Corticosteroids (clobetasol 0.05%) — Patients will receive a maintenance treatment of topical therapy with corticosteroids (clobetasol 0.05%) that will be administered by usual clinical practice.
  Other Names: Control
  Arms: Group Control

SUMMARY:
LIQUENIA clinical trial is a phase II, controlled, prospective and unicentric study to assess vulvar lichen sclerosus (VLS) treatment using adipose tissue associated with autologous platelet-rich plasma (PRP) coming from the inner side of the patients' thighs, which aims to restore the structure and elasticity of the affected vulvar subunits, and to improve vulvar subunits lesions and symptoms, therefore, patients' quality of life from the early phases of the treatment.

DETAILED DESCRIPTION:
Randomized, prospective and unicentric study, in which the investigators evaluate patients with vulvar lichen sclerosus who undergo surgical treatment consisting of two separate infiltrations by intra and subdermal injection in each half vulvar of autologous fatty tissue associated with autologous platelet-rich plasma, in order to:

Main objective:

To estimate the population parameters of the study variables, as well as their variability, to be able to determine the sample size and statistical power for a future clinical trial whose main objective will be to demonstrate the efficacy of this treatment regarding the increase in the vulvar elasticity in patients with vulvar lichen sclerosus.

Secondary Objectives:

1. To evaluate if there is a structural improvement in the vulva areas treated at month, 3 months, 6 months and 12 months after the first infiltration and at 3 and 9 months after the second infiltration.
2. To analysis the improvement of fibrosis and inflammation 6 months after the first infiltration and 3 months after the second infiltration.
3. To study if there is an improvement in symptoms at month, 3 months, 6 months, 12 months after the first infiltration and at 3 months and 9 months after the second infiltration.
4. To examine whether there is an improvement in the quality of patients life.
5. Subsequent use of clinical and pain assessment scale in this study and in another lichen sclerosus vulvar studies with a greater number of patients.
6. To evaluate the adverse events derived from the treatment during the first year after the first infiltration through its registration in the CRD.

ELIGIBILITY:
Inclusion Criteria:

* Adult women between 18 and 70 years old.
* Patients with clear clinical and/or histological diagnosis of vulvar lichen sclerosus (VLS).
* Moderate to severe affectation of the disease at genital level.
* Patients who have taken topical treatment for at least three months with 0.05% clobetasol propionate.
* Prior signed informed consent form.

Exclusion Criteria:

* Pregnant or lactating women.
* Alcoholic patients.
* Patients with malignant disease diagnosed in the last 5 years.
* Patients infected with HSV-II, HPV, HIV, HBV and HCV viruses.
* Injecting drug users.
* Patients with serious active infectious diseases.
* Patients with known allergy or intolerance to any of the aforementioned treatments.
* Patients with inflammatory diseases that may affect the vulvar area (Crohn's disease, ulcerative colitis, psoriasis, eczema).
* Patients with unrealistic expectations regarding the final benefits of the treatment.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Adult women between 18 and 70 years old
Enrollment: 20 (Actual)
Dates: Start 2017-09-06 (Actual); Primary Completion 2019-12-12 (Actual); Study Completion 2019-12-12 (Actual)

PRIMARY OUTCOMES:
Vulvar elasticity measured by the cutometer-dualmpa® | Month 1 after first infiltration.
  Vulvar elasticity will be measured by the cutometer-dualmpa® for the analysis of the elasticity improvement in the plaques of fibrosis at the affected vulvar areas.
Vulvar elasticity measured by the cutometer-dualmpa® | Month 3 after first infiltration.
  Vulvar elasticity will be measured by the cutometer-dualmpa® for the analysis of the elasticity improvement in the plaques of fibrosis at the affected vulvar areas.
Vulvar elasticity measured by the cutometer-dualmpa® | Month 6 after first infiltration.
  Vulvar elasticity will be measured by the cutometer-dualmpa® for the analysis of the elasticity improvement in the plaques of fibrosis at the affected vulvar areas.
Vulvar elasticity measured by the cutometer-dualmpa® | Year 1 after first infiltration.
  Vulvar elasticity will be measured by the cutometer-dualmpa® for the analysis of the elasticity improvement in the plaques of fibrosis at the affected vulvar areas.
Vulvar elasticity measured by the cutometer-dualmpa® | Month 3 after second infiltration.
  Vulvar elasticity will be measured by the cutometer-dualmpa® for the analysis of the elasticity improvement in the plaques of fibrosis at the affected vulvar areas.
Vulvar elasticity measured by the cutometer-dualmpa® | Month 9 after second infiltration.
  Vulvar elasticity will be measured by the cutometer-dualmpa® for the analysis of the elasticity improvement in the plaques of fibrosis at the affected vulvar areas.

SECONDARY OUTCOMES:
Histological improvement measured by the scale for histological assessment. | Month 6
  The histological improvement will be determined in the treatment group by histological comparison of the biopsy samples taken pre-treatment and after 6 months of treatment, and it will be assessed by the evolution of the advanced stages (basal lamina destruction, orthokeratosis, hypergranulocytosis with an infiltrate of lymphocytes and melanophages with Civatte bodies (necrotic keratinocytes) in the papillary dermis) to earlier stages characterized by dermatitis with lymphocytic infiltrate along the epithelial junction.
Improvement in the quality of patients' life measured by skindex-29 questionnaire quality of life. | Month 1, Month 3, Month 6, Year 1
  The skindex-29 is a questionnaire designed for assessing aspects, such as degree of symptoms, psychosocial functioning, and emotional status, for assessing the effects of skin diseases on patient's quality of life.
Improvement in the clinical symptoms by clinical assessment scale. | Month 1, Month 3, Month 6, Year 1
  Clinical assessment scale is a physical examination for current status of the lesions despite treatment with topical corticosteroids. 1 point will be given to the existence of whitish plaques, 2 points to the presence of bruises, hemorrhagic blisters, erosions/ulcers, pain or bleeding during sexual intercourse and 8 points to labial adhesion (minora/major), clítoris phimosis and narrowing of the introitus. The patients with 1 point will be mild patients, the patients with 2-7 points will suffer a moderate affectation while the patients with more than 8 or + points will be in advanced stages with a serious affectation.
Improvement in the pruritus measured by 4D Pruritus Scale. | Month 1, Month 3, Month 6, Year 1
  4D Pruritus Scale is a brief but multidimensional questionnaire to assess itching. The scale scores from 0 (no negative impact) to 4 (greatest negative impact) on pruritus duration, intensity, extent and daily activities disability.
Improvement in the pain measured by Pain Scale. | Month 1, Month 3, Month 6, Year 1
  The pain scale is designed for assessing pain associated with sexual intercourse and urination (2 points), resting and nightime sleep conciliation (6 points).Regarding the gradation of symptoms it will be classified as mild (1 point) the existence of mild pain/discomfort that allows normal life without taking analgesics, moderate (2-5 points) when usual doses of analgesics are required and serious with more than 5 points.
Improvement in sexual performance by Sexual Functioning Index (SFI) | Month 1, Month 3, Month 6, Year 1
  Sexual Functioning Index is a questionnaire related to four topics: sexual activity, sexual intercourse, sexual stimulation and sexual desire.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Gutierrez Ontalvilla, Principal Investigator — Hospital La Fe
Locations (1):
- Hospital Universitario y Politécnico La Fe, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tausch TJ, Peterson AC. Early aggressive treatment of lichen sclerosus may prevent disease progression. J Urol. 2012 Jun;187(6):2101-5. doi: 10.1016/j.juro.2012.01.071. Epub 2012 Apr 12. PMID 22503028
- [Background] Giuseppina Onesti M, Carella S, Ceccarelli S, Marchese C, Scuderi N. The Use of Human Adipose-Derived Stem Cells in the Treatment of Physiological and Pathological Vulvar Dystrophies. Stem Cells Int. 2016;2016:2561461. doi: 10.1155/2016/2561461. Epub 2016 Jan 10. PMID 26880944
- [Background] Boero V, Brambilla M, Sipio E, Liverani CA, Di Martino M, Agnoli B, Libutti G, Cribiu FM, Del Gobbo A, Ragni E, Bolis G. Vulvar lichen sclerosus: A new regenerative approach through fat grafting. Gynecol Oncol. 2015 Dec;139(3):471-5. doi: 10.1016/j.ygyno.2015.10.014. Epub 2015 Oct 21. PMID 26499935
- [Background] Tamburino S, Lombardo GA, Tarico MS, Perrotta RE. The Role of Nanofat Grafting in Vulvar Lichen Sclerosus: A Preliminary Report. Arch Plast Surg. 2016 Jan;43(1):93-5. doi: 10.5999/aps.2016.43.1.93. Epub 2016 Jan 15. No abstract available. PMID 26848453
- [Background] Focseneanu MA, Gupta M, Squires KC, Bayliss SJ, Berk D, Merritt DF. The course of lichen sclerosus diagnosed prior to puberty. J Pediatr Adolesc Gynecol. 2013 Jun;26(3):153-5. doi: 10.1016/j.jpag.2012.12.002. Epub 2013 Mar 16. PMID 23507004
- [Background] Gale KL, Rakha EA, Ball G, Tan VK, McCulley SJ, Macmillan RD. A case-controlled study of the oncologic safety of fat grafting. Plast Reconstr Surg. 2015 May;135(5):1263-1275. doi: 10.1097/PRS.0000000000001151. PMID 25919241
- [Background] Sinno S, Wilson S, Brownstone N, Levine SM. Current Thoughts on Fat Grafting: Using the Evidence to Determine Fact or Fiction. Plast Reconstr Surg. 2016 Mar;137(3):818-824. doi: 10.1097/01.prs.0000479966.52477.8b. PMID 26910662
- [Background] Sehgal VN, Pandhi D, Khurana A. Nonspecific genital ulcers. Clin Dermatol. 2014 Mar-Apr;32(2):259-74. doi: 10.1016/j.clindermatol.2013.08.024. PMID 24559562
- [Background] Fuh KC, Berek JS. Current management of vulvar cancer. Hematol Oncol Clin North Am. 2012 Feb;26(1):45-62. doi: 10.1016/j.hoc.2011.10.006. PMID 22244661
- [Background] Erickson BA, Elliott SP, Myers JB, Voelzke BB, Smith TG 3rd, McClung CD, Alsikafi NF, Vanni AJ, Brant WO, Broghammer JA, Tam CA, Zhao LC, Buckley JC, Breyer BN; Trauma and Urologic Reconstructive Network of Surgeons. Understanding the Relationship between Chronic Systemic Disease and Lichen Sclerosus Urethral Strictures. J Urol. 2016 Feb;195(2):363-8. doi: 10.1016/j.juro.2015.08.096. Epub 2015 Sep 5. PMID 26343349
- [Background] Arrowsmith S, Kendrick A, Wray S. Drugs acting on the pregnant uterus. Obstet Gynaecol Reprod Med. 2010 Aug;20(8):241-247. doi: 10.1016/j.ogrm.2010.05.001. PMID 24443652
- [Background] Brauer M, van Lunsen R, Burger M, Laan E. Motives for Vulvar Surgery of Women with Lichen Sclerosus. J Sex Med. 2015 Dec;12(12):2462-73. doi: 10.1111/jsm.13052. Epub 2015 Nov 27. PMID 26610399
- [Background] Kreuter A, Kryvosheyeva Y, Terras S, Moritz R, Mollenhoff K, Altmeyer P, Scola N, Gambichler T. Association of autoimmune diseases with lichen sclerosus in 532 male and female patients. Acta Derm Venereol. 2013 Mar 27;93(2):238-41. doi: 10.2340/00015555-1512. PMID 23224274
- [Background] Mazzola RF, Mazzola IC. The fascinating history of fat grafting. J Craniofac Surg. 2013 Jul;24(4):1069-71. doi: 10.1097/SCS.0b013e318292c447. No abstract available. PMID 23851740